CLINICAL TRIAL: NCT00563342
Title: Catheters Dysfunction Rate After Instillation of Ethanol 60% Lock Solution in Tunneled Silicone Catheter of Chronic Hemodialysis Patients
Acronym: Ethanol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Bertrand Souweine, CHU Clermont-Ferrand
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CHU-0027
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: End Stage Renal Failure, Hemodialysis
Keywords: Ethanol, lock solution, infection
MeSH Terms: conditions — Renal Insufficiency, Chronic; Infections | interventions — Ethanol

INTERVENTIONS:
Drug: Ethanol — Examine the risk of catheter dysfunction during the dialysis session that follows the instillation of ethanol 60% as lock solution in tunneled silicone catheters of end stage renal failure patients treated by hemodialysis

SUMMARY:
The primary objective of the study is to examine the risk of catheter dysfunction during the dialysis session that follows the instillation of ethanol 60% as lock solution in tunneled silicone catheters of end stage renal failure patients treated by hemodialysis.

The catheters dysfunction rate is the primary outcome. The dysfunction is defined as partial or complete occlusion or infection associated with dialysis catheter.

As a secondary outcome, the dialysis quality is also examined (urea reduction rate, total ultrafiltration)

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, over 18 years,
* Chronic hemodialysis 3 times a week, with two tunnel silicone catheters since at least 15 days,
* Written informed consent
* Social security

Exclusion Criteria:

* Antibiotic therapy during selection phase,
* Partial or complete catheter occlusion during selection phase,
* Venous pressure at dialysis connection > 300 mmHg,
* Known allergy to ethanol,
* Patient involved in any other clinical trial or in the exclusion period
* Severe co-morbidity
* Acute or chronic infectious disease
* Evolutive neoplasia,
* HIV, HCV positive serology at inclusion,
* Scheduled surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The catheters dysfunction rate | as partial or complete occlusion or infection associated with dialysis catheter

SECONDARY OUTCOMES:
The dialysis quality is also examined (urea reduction rate, total ultrafiltration) | as partial or complete occlusion or infection associated with dialysis catheter

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Souweine, Pr, Principal Investigator
Locations (1):
- Lacarin, Clermont-Ferrand, France

REFERENCES:
- [Derived] Coupez E, Timsit JF, Ruckly S, Schwebel C, Gruson D, Canet E, Klouche K, Argaud L, Bohe J, Garrouste-Orgeas M, Mariat C, Vincent F, Cayot S, Cointault O, Lepape A, Darmon M, Boyer A, Azoulay E, Bouadma L, Lautrette A, Souweine B. Guidewire exchange vs new site placement for temporary dialysis catheter insertion in ICU patients: is there a greater risk of colonization or dysfunction? Crit Care. 2016 Jul 30;20(1):230. doi: 10.1186/s13054-016-1402-6. PMID 27473868